CLINICAL TRIAL: NCT03726138
Title: The Association of Sleep and Psychological Symptoms With Prognosis and Onset of MSK Pain; a One-year Prospective Cohort Study in Danish General Practice
Brief Title: The Association of Sleep and Psychological Symptoms With Prognosis of MSK Pain in Danish General Practice
Status: Completed | Type: Observational
Sponsor: Aalborg University (Other)
Collaborators: Research Unit for General Practice in Aalborg (Other)
Responsible Party: Principal Investigator, Sinead Holden, Post- Doctoral Research Fellow, Aalborg University
Other Study IDs: LS MSK FU
Record Dates: First submitted 2018-10-30; First posted 2018-10-31 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2019-01

CONDITIONS: Musculoskeletal Pain; Insomnia; Anxiety; Depressive Symptoms
MeSH Terms: conditions — Musculoskeletal Pain; Sleep Initiation and Maintenance Disorders; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Musculoskeletal (MSK) pain is a major public health concern. Approximately one in four consult their general practitioner (GP) with a musculoskeletal problem during the course of a year, making it the largest diagnostic group.

Modifiable factors including affective disorders (e.g. anxiety and depressive symptoms) and sleep problems may be important prognostic factors for MSK pain. However, there is a lack of prospective research examining the interaction between these conditions in patients with MSK pain in a GP-setting.

DETAILED DESCRIPTION:
This is a prospective cohort study of 299 participants from a GP-setting. Investigators will evaluate the occurrence of MSK pain at one-year follow-up and how the predictors (anxiety, depressive, and sleep problems and multi-site MSK pain) are associated with prognosis of MSK pain.

A secondary aim will be to identify those factors associated with new onset MSK pain. Participants will complete a sleep questionnaire (the ATHENS insomnia questionnaire) containing 8 questions about sleep quality and quantity and a questionnaire (The Hospital Anxiety and Depression Score)) containing 14 questions focusing on anxiety and depression.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 12 years visiting the GP who contributed baseline data and over who consented to be contacted as part of a prospective cohort study

Based on baseline assessment, patients were divided into two separate groups: The MSK pain group and the control group (representing the pain-free background population in general practice).

Inclusion Criteria for MSK pain group:

* Musculoskeletal pain at any body site
* Pain least once a week during the preceding month
* Pain that negatively interfere with the participant's usual activities.

The same criteria for 'MSK pain' apply for the follow-up study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients aged 12 years and over visiting the GP during the study period in November 2017. The patients who consented to participate in the follow-up (299 patients) are eligible for one-year follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Musculoskeletal pain (persistence) | 1 year
  The primary outcome of this study will be MSK pain as evaluated by a self-report pain questionnaire. To be classified as having MSK pain, the pain must occur at least weekly and negatively interfere with the patient's usual activities. The prevalence of MSK pain at follow-up will be assessed to determine if patients from general practice who reported MSK pain at baseline still have MSK pain at one-year follow-up

SECONDARY OUTCOMES:
New onset musculoskeletal pain | 1 year
  This outcome will be new onset MSK pain assessed by a self-report pain questionnaire. The incidence of MSK pain at one-year follow-up will be assessed among patients from general practice who reported no MSK pain at baseline.
  To be classified as having MSK pain, the pain must occur at least weekly and negatively interfere with the patient's usual activities.

CONTACTS AND LOCATIONS:
Overall Officials: Sinead Holden, PhD, Principal Investigator — Research Unit for General Practice in Aalborg
Locations (1):
- Research Unit for General Practice in Aalborg, Aalborg, Denmark